CLINICAL TRIAL: NCT06292442
Title: Effects of High-Intensity Interval Training on Muscle Strength, Atrophy and Aerobic Capacity in Stroke Patients.
Brief Title: Effects of HIIT on Muscle Strength, Atrophy and Aerobic Capacity in Stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0237
Record Dates: First submitted 2024-01-28; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Stroke
Keywords: aerobic capacity, chronic stroke, high-intensity interval training, muscle atrophy, muscle strength, stroke
MeSH Terms: conditions — Stroke; Muscular Atrophy | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional physical therapy (Active Comparator): This group received conventional physical therapy treatment including Range of Motion (ROM) exercises for the affected hip, knee, and ankle joints, as well as stretching exercises for tight lower limb muscles, administered 3 times per week for 4 weeks, with each session lasting approximately 20-30 minutes.
  Interventions: Other: traditional physical therapy
- High intensity interval training (Experimental): This group received high-intensity interval training along with conventional treatment for the lower limb muscles
  Interventions: Other: High intensity interval training

INTERVENTIONS:
Other: traditional physical therapy — This group received conventional physical therapy treatment including Range of Motion (ROM) exercises for the affected hip, knee, and ankle joints, as well as stretching exercises for tight lower limb muscles, administered 3 times per week for 4 weeks, with each session lasting approximately 20-30 minutes.
  Arms: Traditional physical therapy
Other: High intensity interval training — This group received High Intensity interval training along with conventional treatment for lower limb muscles, performed 3 times per week fr 4 weeks.
  Arms: High intensity interval training

SUMMARY:
To determine the effects of High-Intensity Interval Training on muscle strength, atrophy, and aerobic capacity in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females were included
* aged 40-60 years
* Chronic stroke patients who experienced a first-ever ischemic stroke
* Stable cardiovascular condition (American Heart Association class B)
* Physician clearance to participate in a 4-week HIIT program
* No prior structured exercise in the last 3 months
* Ability to walk 10 m over ground with or without assistive devices
* Patients who scored >24/30 on MMSE (Mini-Mental State Examination)

Exclusion Criteria:

* Patients who were hospitalized for cardiac or pulmonary disease within the past 3 months
* Patients who had implanted pacemaker or defibrillator
* Patients having conditions where VO2peak assessment is contraindicated, such as uncontrolled hypertension(>180/100), severe aortic stenosis, acute myocarditis, recent myocardial infarction, or other acute cardiovascular events within the past three months, were excluded from the study
* Patients with severe lower limb spasticity (Ashworth Scale scores >2 of 4 for knee flexion, knee extension, or ankle dorsiflexion)
* Pregnant females
* Previous exposure to fast treadmill walking in the past year

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 4th week
  Manual Muscle Testing is a test that is used to assess muscle strength.
Muscle Atrophy | 4th week
  Measuring tape is used to measure the calf circumference to measure the atrophy, muscle size over time.
6-Minute Walk Test (6MWT) | 4th week
  6-Minute Walk Test (6MWT) used to measure Functional capacity, aerobic fitness and endurance.
Aerobic Capacity | 4th week
  Harvard Step Test is used to measure Functional capacity, aerobic fitness and endurance.

SECONDARY OUTCOMES:
Fastest Gait Speed | 4th week
  10-Meter Walk Test is a test used for assessing gait speed, monitoring rehabilitation progress, functional assessment, fall risk assessment, and research purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah international university lahore campus
Locations (1):
- Jinnah Hospital, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hugues N, Pellegrino C, Rivera C, Berton E, Pin-Barre C, Laurin J. Is High-Intensity Interval Training Suitable to Promote Neuroplasticity and Cognitive Functions after Stroke? Int J Mol Sci. 2021 Mar 16;22(6):3003. doi: 10.3390/ijms22063003. PMID 33809413
- [Background] Gjellesvik TI, Becker F, Tjonna AE, Indredavik B, Lundgaard E, Solbakken H, Brurok B, Torhaug T, Lydersen S, Askim T. Effects of High-Intensity Interval Training After Stroke (The HIIT Stroke Study) on Physical and Cognitive Function: A Multicenter Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 Sep;102(9):1683-1691. doi: 10.1016/j.apmr.2021.05.008. Epub 2021 Jun 6. PMID 34102144
- [Background] Krawcyk RS, Vinther A, Petersen NC, Faber J, Iversen HK, Christensen T, Klausen TW, Kruuse C. High-intensity training in patients with lacunar stroke: A one-year follow-up. J Stroke Cerebrovasc Dis. 2023 Apr;32(4):106973. doi: 10.1016/j.jstrokecerebrovasdis.2022.106973. Epub 2023 Jan 7. PMID 36623990
- [Background] Boyne P, Billinger SA, Reisman DS, Awosika OO, Buckley S, Burson J, Carl D, DeLange M, Doren S, Earnest M, Gerson M, Henry M, Horning A, Khoury JC, Kissela BM, Laughlin A, McCartney K, McQuaid T, Miller A, Moores A, Palmer JA, Sucharew H, Thompson ED, Wagner E, Ward J, Wasik EP, Whitaker AA, Wright H, Dunning K. Optimal Intensity and Duration of Walking Rehabilitation in Patients With Chronic Stroke: A Randomized Clinical Trial. JAMA Neurol. 2023 Apr 1;80(4):342-351. doi: 10.1001/jamaneurol.2023.0033. PMID 36822187
- [Background] Miller A, Reisman DS, Billinger SA, Dunning K, Doren S, Ward J, Wright H, Wagner E, Carl D, Gerson M, Awosika O, Khoury J, Kissela B, Boyne P. Moderate-intensity exercise versus high-intensity interval training to recover walking post-stroke: protocol for a randomized controlled trial. Trials. 2021 Jul 16;22(1):457. doi: 10.1186/s13063-021-05419-x. PMID 34271979
- [Background] Anjos JM, Neto MG, Dos Santos FS, Almeida KO, Bocchi EA, Lima Bitar YS, Duraes AR. The impact Of high-intensity interval training On functioning And health-related quality Of life In post-stroke patients: A systematic review With meta-analysis. Clin Rehabil. 2022 Jun;36(6):726-739. doi: 10.1177/02692155221087082. Epub 2022 Mar 15. PMID 35290104
- [Background] Boyne P, Miller A, Schwab SM, Sucharew H, Carl D, Billinger SA, Reisman DS. Training parameters and longitudinal adaptations that most strongly mediate walking capacity gains from high-intensity interval training post-stroke. medRxiv [Preprint]. 2023 Feb 23:2023.02.20.23286194. doi: 10.1101/2023.02.20.23286194. PMID 36865178
- [Background] Hsu CC, Fu TC, Huang SC, Chen CP, Wang JS. Increased serum brain-derived neurotrophic factor with high-intensity interval training in stroke patients: A randomized controlled trial. Ann Phys Rehabil Med. 2021 Jul;64(4):101385. doi: 10.1016/j.rehab.2020.03.010. Epub 2020 May 11. PMID 32344098
- [Background] Boyne P, Doren S, Scholl V, Staggs E, Whitesel D, Carl D, Shatz R, Sawyer R, Awosika OO, Reisman DS, Billinger SA, Kissela B, Vannest J, Dunning K. Preliminary Outcomes of Combined Treadmill and Overground High-Intensity Interval Training in Ambulatory Chronic Stroke. Front Neurol. 2022 Feb 4;13:812875. doi: 10.3389/fneur.2022.812875. eCollection 2022. PMID 35185766
- [Background] Plummer P. Critically appraised paper: High-intensity interval training after stroke improves some aspects of physical function, but benefits are not sustained. J Physiother. 2022 Jul;68(3):204. doi: 10.1016/j.jphys.2022.05.014. Epub 2022 Jun 14. No abstract available. PMID 35715374